CLINICAL TRIAL: NCT01193595
Title: An Open-label, Non-randomized, Dose Escalation, Safety and Pharmacokinetic Phase I Study of Ombrabulin (AVE8062) in Combination With Bevacizumab Administered by Intravenous Infusion Every 3 Weeks in Patients With Advanced Solid Tumors.
Brief Title: Dose-escalation, Safety, Pharmacokinetics Study of AVE8062 Combined With Bevacizumab in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCD11379; 2009-017797-20 (EudraCT Number)
Record Dates: First submitted 2010-08-31; First posted 2010-09-02 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Neoplasms, Malignant
MeSH Terms: conditions — Neoplasms | interventions — AC 7700; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AVE8062/ bevacizumab (Experimental): The combination of ombrabulin and bevacizumab will be administered every 3 weeks according to the following schedule: One day 1, ombrabulin will be administered as a 30 minutes intravenous (i.v) infusion. Bevacizumab will be administered as a 30-90 minutes i.v. infusion 24 hours after the end of ombrabulin infusion on day 2.
  Interventions: Drug: Ombrabulin (AVE8062); Drug: bevacizumab

INTERVENTIONS:
Drug: Ombrabulin (AVE8062) — Pharmaceutical form:Solution for infusion
  Route of administration: Intravenous
Drug: bevacizumab — Pharmaceutical form:Solution for infusion
  Route of administration: Intravenous

SUMMARY:
Primary Objective:

- To determine the maximum administered dose (MAD) and the maximum tolerated dose (MTD) of ombrabulin in combination with best tolerated dose of bevacizumab based on the incidence of related Dose Limiting Toxicities (DLTs).

Secondary Objectives:

* To assess the overall safety profile of the combination
* To characterize the pharmacokinetic (PK) profile of both ombrabulin and bevacizumab when given in combination
* To evaluate preliminary evidence of anti-tumor activity
* To assess the pharmacodynamic effect using (Dynamic Contrast Enhanced Ultra-Sound) DCE-US, measuring biomarkers

DETAILED DESCRIPTION:
The duration of the study for each patient will include an up to 28-day screening phase, 21-day study treatment cycles, an end of treatment visit with a follow-up period. Each patient will participate in only one dose group and will receive AVE8062 with bevacizumab every 3 weeks until disease progression or unacceptable toxicities, withdrawal of consent or Investigator's decision.

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically proven solid malignant tumor at the first diagnosis with the exception of squamous non small cell lung cancer (NSCLC).
* Advanced neoplastic disease (i.e. metastatic or locally unresectable advanced disease)
* Presence of one measurable lesion at baseline in the MTD expanded cohort

Exclusion criteria:

* ECOG (Eastern cooperativeOncology Group) performance status > 1
* Concurrent treatment with any other anticancer therapy
* Pericardial effusion requiring intervention (drainage)
* History of brain metastasis, spinal cord compression or carcinomatous meningitis or new evidence of brain metastasis on screening Computed tomography (CT) or Magnetic resonance imaging (MRI) scan
* Diagnosis of squamous Non Squamous Cell Lung Cancer (NSCLC) or with mixed cell type with predominant squamocellular histology
* Hormone sensitive prostate cancer
* Abdominal Radiotherapy
* Major surgery within the last month of study enrollment or surgical wound not fully healed before study enrollment
* High cumulative doses of anthracycline
* Inadequate organ function
* Inadequate hematology function or poor bone marrow reserve
* Any of the following within 6 months prior to study enrollment: peptic ulcer disease, erosive oesophagitis or gastritis, infectious or inflammatory bowel disease and diverticulitis
* Any history or underlying cardiac condition that may increase the risks associated with the study participation or administration of the investigational products, or that may interfere with the interpretation of the results.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) that will define the MTD | 3 weeks

SECONDARY OUTCOMES:
Overall safety profile of the combination | up to a maximum follow-up of 1 year
Pharmacokinetic parameters of ombrabulin | 6 weeks
Pharmacokinetic parameters of bevacizumab | 6 weeks
Preliminary evidence of antitumor activity according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) | up to a maximum follow-up of 1 year
Pharmacodynamic effect (biomarkers) | cycle 1

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (4):
- Investigational Site Number 250001, Villejuif, France
- Italy (2):
  - Investigational Site Number 380002, Milan
  - Investigational Site Number 380001, Milan
- Investigational Site Number 826001, Sutton, United Kingdom